# Statistical Analysis Plan

Study Title: The effects of PF-04995274 on emotional processing in treatment-resistant, medicated, depressed patients (RESTART study).

CT REGISTRATION: NCT03515733. ETHICS REF: 18/SC/0074

#### **Objectives**

The primary aim of the study is to investigate the effects of 7 days of PF-04995274 administration (adjunctive to SSRI/SNRI medication) on behavioural measures of non-emotional and emotional cognition, specifically memory performance on an auditory verbal learning task and performance (including accuracy and reaction times) on a facial expression recognition task. The secondary aim of the study is to investigate the effects of 7 days of PF-04995274 administration (adjunctive to SSRI/SNRI medication) on other behavioural measures of non-emotional and emotional cognition.

#### Brief summary of design

This study uses a double-blind, placebo-controlled, randomised between-groups design. Participants are patients who fulfil criteria for current episode of Major Depressive Disorder (MDD) and are currently taking an SSRI/SNRI and have failed to response clinically. Participants will be randomised to receive 7-9 days treatment with either PF-04995274 (15 mg daily) or a matched placebo. This study includes three visits in total: (a) Screening Visit; (b) First Dose Visit; (c) Research Visit Two. All visits will take place at the Warneford Hospital, Oxford University Department of Psychiatry.

#### **Determination of Sample Size**

We will recruit 50 participants to the study (25 on PF-0499574 and 25 on placebo). Participants who withdraw during the study or do not provide complete data-sets will be replaced. Based on data acquired in Harmer et al., (2004) comparing citalopram to placebo, if we aim for 0.9 power and a 0.05 false positive rate, a suggested group sample size is 19 (G\*power) to ensure determination of group level differences at this variable if they exist. As 5HT4 agonism is less well studied, and to account for the exclusion of low quality data before analysis, we will aim for 25 individuals with complete datasets per group (total sample size of 50).

#### **Data Cleaning**

- Will be performed prior to unblinding
- Outliers will be excluded on a per task basis
- For all behavioural data, excluding the EPS, cut-off thresholds will be determined based on a visual inspection of a histogram plot, examining thresholds for:
  - > Trials with unusually low response times
  - > Trials with unusually high response times
  - Proportion of missing/removed trials per participant
  - Abnormally low mean accuracy (or equivalent outcome) per participant
  - Abnormally high mean reaction time per participant
- For all self-report data, extreme outliers indicating invalid data entry will be determined based on a visual inspection of a histogram plot
- For emotion potentiated startle data, two researchers will independently a) distinguish startle blink response from noise and decide whether a response could have been seen, had one occurred, excluding trials if no response could not be seen and b) determine if there is a blink response or if the trial should be recorded as a non-response. If there is disagreement, a third researcher will make a final decision.

## Behavioural Analysis

Below is a non-exhaustive list of outcomes and analyses which will be conducted.

| Behavioural Task | Outcomes | Analysis |
|---|---|---|
| | | <ul> <li>All key endpoints will be summarized (mean, standard deviation) in<br/>tables and bar charts (mean ±SEM)</li> </ul> |
| | | Conducted in R (version will be confirmed in publications) |
| Facial Expression | Unbiased hit rate, as described by Wagner (1993) – a | Repeated measures analyses of variance (ANOVAs): |
| Recognition Task (FERT) | measure of emotion identification accuracy which | Between-subject factor – 2 levels: Treatment group (PF- |
| | accounts for response bias i.e. any general tendency to | 04995274 or placebo) |
| Recognition of computer- | identify the emotion when it is not present. Calculated as | Within-subject factor – 7 levels (Fear, anger, happy, surprise, |
| based positive and negative | proportion of correct hits * (number of hits/all hits and | disgust, sad, neutral) |
| facial expressions | misses), for each facial expression category. | |
| | % correct and response bias will also be reported | |
| P1vital® Limited Products | individually. | |
| | Misclassifications: Number of responses to each facial | |
| | expression category incorrectly classified as another facial | |
| | expression category e.g. identifying a fearful face as | |
| | surprised | |
| | Reaction time (ms) for trials with correct responses. | |
| Auditory Verbal Learning | Number of words recalled - | Repeated measures analyses of variance (ANOVAs): |
| Task (AVLT) | List A immediate recall trials | <ul> <li>Between-subject factor – 2 levels: Treatment group (PF-<br/>04995274 or placebo)</li> </ul> |
| Recall of words read aloud | | Within-subject factor - 5 levels (List A immediate recall trials 1-5) |

| Pen and paper | Number of words recalled - | Repeated measures analyses of variance (ANOVAs): |
|---|---|---|
| | List A short delay | Between-subject factor – 2 levels: Treatment group (PF- |
| | Number of words recalled - | 04995274 or placebo) |
| | List A long delay | Within-subject factor - 2 levels (List A short and long delay |
| | | trials) |
| | Number of intrusions (words incorrectly recalled) across | Independent samples t-tests |
| | List A acquisition trials | |
| | Number of repetitions (words repeated within the same | |
| | trial) across List A acquisition trials | |
| | Number of words recalled - | |
| | List B recall | |
| | Number of hits and false alarms in the delayed | |
| | recognition test | |
| Probabilistic Instrumental | % Accuracy (correct or incorrect symbol choice) | Independent samples t-tests |
| Learning Task (PILT) | Correct = symbol associated with high probability of | |
| | winning or low probability of losing | |
| Reward sensitivity | Proportion of group choosing correct symbol per trial | The proportion will be calculated, and plotted on a learning curve |
| | | to determine where learning plateaus. |
| Neurobehavioral Systems | | |
| Presentation software | | Repeated measures analyses of variance (ANOVAs) - trials where |
| (https://www.neurobs.com) | | learning has plateaued |
| | | Between-subject factor – 2 levels: Treatment group (PF- |
| | | 04995274 or placebo) |
| | | Within-subject factor – 2 levels: Condition (win or loss) |
| | Learning rate from reinforcement learning model | Repeated measures analyses of variance (ANOVAs) |
| | | Between-subject factor – 2 levels: Treatment group (PF- |
| | | 04995274 or placebo) |
| | | Within-subject factor – 2 levels: Condition (win or loss) |

| | Decision temperature parameters from reinforcement learning model Amount won Amount lost Total monetary amount earned | Repeated measures analyses of variance (ANOVAs) • Between-subject factor – 2 levels: Treatment group (PF-04995274 or placebo) • Within-subject factor – 2 levels: Condition (win or loss) Independent samples t-tests |
|---|---|---|
| Emotional Categorisation Task (ECAT) Categorisation of emotional words | % Accuracy – words correctly identified as positive or negative | <ul> <li>Mixed model analyses of variance (ANOVAs).</li> <li>Between-subject factor – 2 levels: Treatment group (PF-04995274 or placebo)</li> <li>Within-subject factor – 2 levels: Word valence (positive or negative)</li> </ul> |
| P1vital® Limited Products Emotional Recall Task (EREC) Recall of emotional words from ECAT | Reaction time Number of hits (words recalled correctly) Number of false alarms (words recalled incorrectly) | - |
| P1vital® Limited Products Emotional Recognition Task (EMEM) | Number of hits (words recognised correctly) Number of false alarms (words recognised incorrectly) | |
| Recognition of emotional words from ECAT P1vital® Limited Products | Reaction time | |

| Facial Dot Probe Task | Vigilance scores derived from reaction time – e.g. bias | Mixed models analyses of variance (ANOVAs). |
|---|---|---|
| (FDOT) Vigilance to fearful and happy faces P1vital® Limited Products | scores calculated by subtracting median reaction times in congruent trials (i.e. the probe appears behind the emotional expression) from those in incongruent trials (i.e. the probe appears behind the neutral expression) | <ul> <li>Between-subject factor – 2 levels: Treatment group (PF-04995274 or placebo)</li> <li>Within-subject factors <ul> <li>2 levels: Emotion (positive or negative)</li> <li>2 levels: Probe duration (masked or unmasked)</li> </ul> </li> </ul> |
| Emotion Potentiated | Raw amplitude of startle response | Mixed models analyses of variance (ANOVAs). |
| Startle (EPS) | Raw amplitude of startle response | Between-subject factor – 2 levels: Treatment group (PF-<br>04995274 or placebo) |
| EMG data, in response to white noise during positive or negative images | Z-transformed amplitude of startle response | <ul> <li>Within-subject factors – 2 levels: Trial type (positive, negative, neutral)</li> </ul> |
| San Diego Instruments, San<br>Diego, CA, USA | Latency of startle response (ms) | |
| Oxford Memory Test<br>(OMT) | Proportion of correct probe selections | Mixed models analyses of variance (ANOVAs). Between-subject factor – 2 levels: Treatment group (PF- |
| Visual short term spatial memory | Absolute error for probe location Reaction Time | <ul> <li>04995274 or placebo)</li> <li>Within-subject factors – 2 levels: Trial condition (1 or 3 memory probes)</li> </ul> |
| Oxford Memory Test application "Short_Fractals1" — modified from "What was where task" (Pertzov et al., 2013) running on iOS 12.3.1 | | |

| Self-report or researcher-observed scale – all completed on Qualtrics.XM (https://www.qualtrics.com) except HAM-D | | |
|---|---|---|
| Eysenck Personality Questionnaire (EPQ) | Total score for each dimension | Report descriptives for each group |
| State and Trait Anxiety Inventory – | Total score | |
| Trait subscale (STAI-T) | | |
| Becks Depression Inventory (BDI) | Total score | |
| Hamilton Depression Scale (HAM-D) | Total score | |
| Pen and paper – scored by research team | | |
| Snaith-Hamilton Pleasure Scale (SHAPS) | Total score | |
| State and Trait Anxiety Inventory – | Total score | Mixed model ANOVAs: |
| State subscale (STAI-S) | | Between-subject factor – 2 levels: Treatment group (PF-04995274 or |
| Positive and Negative Affect Scale | Total score for positive and negative | placebo) |
| (PANAS) | subscales | • Within-subject factors – 4 levels: Time condition (Pre-scan, Post-scan, |
| Visual Analogue Scales (VAS) | Total score for each VAS (happy, sad, hostile, alert, anxious, calm) | Pre-ETB, Post-ETB) |
| Side effects | Presence of side effect Severity of side effect Belief in relationship to drug | Descriptive report of frequency of side-effects for each group at four time points (baseline, pre-dose, post-dose and all other study days combined). |
| | | A generalised linear model will be used to analyse side effects, with presence of side-effect as outcome and predictors including treatment group (PF-04995274 or placebo) and time point (baseline, pre-dose, post-dose, day 2/3/4/5/6/7/8/9). |
| | | For side effects significantly associated with group and time-point, we will investigate severity and belief in relationship to study drug. |

When conducting ANOVAs, the Greenhouse-Geisser procedure will be used to correct the degrees of freedom where assumptions of equality of variance are violated. If there is a significant group x condition interaction found in ANOVAs. Post hoc independent samples t tests will be performed to follow up any significant interactions. We will not use the Bonferroni correction for multiple comparisons for post-hoc tests. When conducting t tests, degrees of freedom will be corrected where the assumption of equal variances between groups is violated (i.e. Levene's Test is significant).

### Record of version changes and unblinding

| Date | Version | Blinding Status | Comments |
|---|---|---|---|
| 28 <sup>th</sup> October 2022 | 1.0 | Team blinded, barring unblinding for study medics (AdeC, PC and BG) where necessary. | Data collection complete. First version of complete stats plans. Uploaded to clinicaltrials.gov and OSF. |

#### Study Team involved in analysis

AdeC - Dr Angharad de Cates - DPhil Student, Study Medic

AG - Dr Amy Gillespie – Post-doctoral Researcher

BG - Dr Beata Godlewska - Study Medic

CH - Professor Catherine Harmer - Principal Investigator

MB - Merethe Blandhol - Research Assistant

PC - Professor Phil Cowen – Principal Investigator, Study Medic

SM - Dr Susannah Murphy - Senior Research Fellow